CLINICAL TRIAL: NCT06502509
Title: How Does Kombucha Tea Improve Difficulty During Defecation in Patients With Schizophrenia- A Randomized, Double-blinded, Placebo-controlled, Parallel Study
Brief Title: Kombucha Tea for Improving Defecation in Patients With Schizophrenia- a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Collaborators: CHYUAN JEOU RONG ENTERPRISE CO., LTD (Unknown)
Responsible Party: Principal Investigator, An-Yu Hong, Doctor, TsaoTun Psychiatric Center, Department of Health, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TTPC-113015
Record Dates: First submitted 2024-02-07; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Constipation; Kombucha Tea
MeSH Terms: conditions — Schizophrenia; Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Lemon kombucha tea) arm (Active Comparator)
  Interventions: Dietary Supplement: Commercial Kombucha tea (Brand name E-Ben Organic Kombucha Lemon)
- controlled (Lemon tea) arm (Placebo Comparator)
  Interventions: Dietary Supplement: Lemon tea

INTERVENTIONS:
Dietary Supplement: Commercial Kombucha tea (Brand name E-Ben Organic Kombucha Lemon) — Commercial lemon kombucha tea (Brand:E-Ben Organic Kombucha Lemon), which will be given to participants in opaque bottles for 8 weeks.
  Arms: interventional (Lemon kombucha tea) arm
Dietary Supplement: Lemon tea — Diluted lemon juice with the same pH as the commercial kombucha tea as placebo, which will be given to participants in opaque bottles for 8 weeks.
  Arms: controlled (Lemon tea) arm

SUMMARY:
Patients with schizophrenia frequently have difficulties in bowel habits due to medical adverse effects and unhealthy lifestyle, and the use of various interventions to ameliorate the problems have been noted in clinical setting. Probiotics including Kombucha tea have been proved to modulate the human gut microbiota which may help to improve the stool passage, and have been attracting the public attention across the world. However, little is known among the patients with schizophrenia. In the present study, the research team intends to evaluate effectiveness of Kombucha tea when used in the clinical settings.

ELIGIBILITY:
* Inclusion Criteria:

  1. Inpatient patients diagnosed of schizophrenia according to DSM-5 criteria with the ICD-10-CM codes of F20.x. and hold the cards for Severe Illness issued by the National Health Insurance Administration, and
  2. Are currently and have been hospitalized at the psychiatric rehabilitation ward for more than 6 months, and
  3. Are at relatively stable psychiatric state and able to clearly express their perception or observed bowel conditions, and
  4. Are able to read or communicate with Mandarin or Taiwanese, and
  5. Are able to consent the agreements, and
  6. Subjectively experience difficulty in stool passage, such as decreased frequency, requiring medication or mechanic aids for defecating.
* Exclusion Criteria:

  1. Having an allergic history to fermented food, alcohol or other food, or 2. Severely impaired in cognitive performance, or 3. Having medications, antibiotics, probiotic or other fermented products that may influence gut microbiota at the time or within 3 months of the study, or 4. Having the illness that may affect stool passage or related with intestinal obstruction, such as severe gut disease, intestinal incarceration, tumor, inflammation, stenosis, or hemorrhoid, or 5. Having received major gastro-intestinal surgeries, or 6. Having the ongoing or history of medical illnesses, such as cancers, chronic obstructive pulmonary diseases, peripheral vascular diseases, autoimmune diseases, chronic kidney diseases, diseases involving abnormal metabolic function of visceral organs, or current infections, or 7. Participating other ongoing interventional research that may interfere the implementation or the results of present studies, or 8. Being obviously unable to comply with the execution of the study, or 10. Being declared of guardianship.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
The subjective amelioration of stool passage | The subjective main outcome will be assessed weekly for 12 weeks.
  The subjective amelioration of stool passage: the participants' perceived overall ease of feces on a VAS scale.
The objective amelioration of stool passage | The objective outcome will be assessed at baseline, week 4, 8 and 12 (endpoint).
  The objective amelioration of stool passage: the frequency or the amount of laxative agent use recorded in clinical care.

SECONDARY OUTCOMES:
Adverse effects Adverse effects Adverse effects Adverse effects | Adverse effects will be assessed weekly from Week 1 to Week 12.
  Adverse effects will be assessed by the investigators with a prepared checklist developed by the research team based on the NIH Adverse Event Data Preparation Checklist and the discomforts commonly reported by the Kombucha tea drinkers from literature search.
Stool form | Stool form will be assessed daily from Week 1 to Week 12.
  Stool form will be assessed with the Bristol Stool Form Scale (BSFS) by the participants' reports.
The participants' perceived flatulence, ease and frequency of stool passage. | The participants' perceived flatulence, ease and frequency of stool passage will be assessed weekly from Week 1 to Week 12.
  The participants' perceived flatulence, ease and frequency of stool passage will be assessed on a VAS scale.

OTHER OUTCOMES:
Demographic data | Demographic data will be assessed at baseline.
  Demographic data including sex, body metrics, past medical and allergic history, and other information related with this study will be assessed by research assistants.
Medication list | Medication list of the participants will be assessed at baseline, Week 4, Week 8 and the endpoint (Week 12).
  Medication list of the participants will be obtained and assessed by research pharmacists, and all the medications will be recorded and categorized according to the anatomical therapeutic chemical (ATC) classification. The defined daily dose (DDD) of psychotropic and laxative agents will specifically be calculated.
Psychiatric condition | Psychiatric condition will be assessed at baseline, Week 8 and Week 12.
  Psychiatric condition will be assessed with brief psychiatric rating scale (BPRS) by psychiatrists.
Cognitive condition | Cognitive condition will be assessed at baseline, Week 8 and Week 12.
  Cognitive condition will be assessed with Montreal cognitive assessment (MoCA) by clinical psychologists.
Level of physical activity | Level of physical activity will be assessed at baseline, Week 8 and Week 12.
  Level of physical activity will be assessed according to metabolic equivalents (METs) by occupational therapists.

CONTACTS AND LOCATIONS:
Overall Officials: An-Yu Hong, Principal Investigator — Tsao-Tun Psychiatric Center, Ministry of Health and Welfare; Ying-Jyun Shih, Principal Investigator — Tsao-Tun Psychiatric Center, Ministry of Health and Welfare
Locations (1):
- Tsao-Tun Psychiatric Center, Caotun, Taiwan